CLINICAL TRIAL: NCT06966349
Title: Quantifying Ocular Surface Aberrations After Tear Film Interventions
Acronym: GAMBIA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Waterloo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 47100
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-09

CONDITIONS: Tear Film Characteristics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Experimental: Systane Complete / Senofilcon A/ Somofilcon A (Experimental): On the first day of the study, one drop of Systane Complete will be instilled in each eye. On the second day of the study, senofilcon A will be worn in both eyes. On the third day of the study, somofilcon A will be worn in both eyes.
  Interventions: Drug: Systane Complete Preservative-Free; Device: Senofilcon A; Device: Somofilcon A
- Experimental: Systane Complete/ Somofilcon A/ Senofilcon A (Experimental): On the first day of the study, one drop of Systane Complete will be instilled in each eye. On the second day of the study, somofilcon A will be worn in both eyes. On the third day of the study, senofilcon A will be worn in both eyes.
  Interventions: Drug: Systane Complete Preservative-Free; Device: Senofilcon A; Device: Somofilcon A

INTERVENTIONS:
Drug: Systane Complete Preservative-Free — One drop of Systane Complete Preservative Free will be instilled in each eye.
  Higher order aberrations assessed before and after instillation.
Device: Senofilcon A — Daily disposable silicone hydrogel contact lenses indicated for myopia or hyperopia.
  Higher order aberrations assessed before and after instillation.
  Other Names: ACUVUE OASYS MAX 1-Day
Device: Somofilcon A — Daily disposable silicone hydrogel contact lenses indicated for myopia or hyperopia.
  Higher order aberrations assessed before and after instillation.
  Other Names: clariti 1 day

SUMMARY:
The CA-800 Corneal Analyzer (Visia Imaging S.R.L., Italy) is a device that can measure small imperfections in the tear film when the eyes are open. The goal of this study is to see if the device can detect changes in the tear film after instillation of an eye drop or when contact lenses are worn.

ELIGIBILITY:
Inclusion Criteria:

1. Are at least 17 years of age and have full legal capacity to volunteer.
2. Have signed the information consent letter.
3. Are willing and able to follow instructions and maintain the appointment schedule.
4. Habitually wear spherical soft contact lenses (no multifocal lens, no toric lens wear or extended (overnight) wear).
5. Have a vertex-corrected refractive astigmatism of no more than 0.75D in each eye.
6. Achieve a best corrected visual acuity of 0.00 logMAR or better in each eye.
7. Agree to wear the study contact lenses for at least 6 hours.
8. Have clear corneas (e.g. no central scars).
9. Have no active ocular disease or inflammation.

Exclusion Criteria:

1. Are participating in another concurrent clinical research study.
2. Have worn any rigid contact lenses in the past 30 days.
3. Have been diagnosed with irregular cornea (e.g., keratoconus, etc.).
4. Have any known active ocular condition, disease, and/or infection.*
5. Have a systemic or ocular condition that, in the opinion of the investigator, may affect a study outcome variable.
6. Have a known sensitivity to the diagnostic sodium fluorescein to be used in the study.
7. Have undergone refractive error surgery.
8. Are a member of the study team for this study, i.e. are listed on the delegation log for this study.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in higher order aberrations with an eye drop | Baseline (prior to instillation); immediately, 10, 20, 30, and 60 minutes post instillation of an eye drop
  The change in root mean square (measured in microns) was assessed over 20 seconds. Data from the right eye was analyzed.
Change in higher order aberrations with senofilcon A | Baseline (prior to insertion); immediately, 30 minutes, and 6 hours post insertion of a contact lens
  The change in root mean square (measured in microns) was assessed over 20 seconds. Data from the right eye was analyzed.
Change in higher order aberrations with somofilcon A | Baseline (prior to insertion); immediately, 30 minutes, and 6 hours post insertion of a contact lens
  The change in root mean square (measured in microns) was assessed over 20 seconds. Data from the right eye was analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD, DSc, FCOptom, Principal Investigator — Centre for Ocular Research & Education
Locations (1):
- Centre for Ocular Research & Education, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No